CLINICAL TRIAL: NCT03508089
Title: Exploration of Microcirculatory Alteration and Endothelial Dysfunction by Adaptive Optics in Multiple Sclerosis
Acronym: MS-EYE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Dr Dan BUCH, Principal Investigator, Versailles Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P15/18_ MS-EYE
Record Dates: First submitted 2018-03-25; First posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Sclerosis, Multiple
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Other)
  Interventions: Other: Ocular Fundus on voluntary person
- Multiple Sclerosis Arm (Active Comparator)
  Interventions: Other: Ocular fundus on patient with Multiple Sclerosis

INTERVENTIONS:
Other: Ocular fundus on patient with Multiple Sclerosis — Ocular fundus on patient with Multiple Sclerosis
  Arms: Multiple Sclerosis Arm
Other: Ocular Fundus on voluntary person — Ocular Fundus on voluntary person
  Arms: Control Arm

SUMMARY:
It's a pilot, interventional prospective monocentric study. It aims to compare the wall / lumen ratio (WLR) of retinal arterioles (common marker of microangiopathies) between patients with multiple sclerosis and controls using the technique of adaptive optics.

ELIGIBILITY:
Patient Inclusion Criteria

* Major patient between 18 and 50 years
* Patient with relapsing or remitting multiple sclerosis defined according to revised Mc Donald criteria 2010
* Written, free and informed consent dated and signed
* Patient affiliated to a social security scheme

Control Inclusion Criteria:

* Person between the ages of 18 and 50
* Written, free and informed consent dated and signed
* Person affiliated to a social security scheme
* Person with multiple sclerosis

Exclusion Criteria:

* Contraindication to the use oxygen (O2): Acute or chronic respiratory insufficiency
* Pregnant or lactating woman
* Inability to see fundus (cataract), retinopathy, glaucoma
* Use of vasoactive substances (eg nasal decongestants, triptans, alkaloids) in the last 48 hours
* Use of nonsteroidal anti-inflammatory drugs (ibuprofen, naproxen, ..) and steroids (corticosteroids) in the last 48 hours
* Known Diabetes or taking antidiabetics in the last 48 hours
* Use of statins in the last 48 hours
* Known hypertension or antihypertensive treatment in the last 48 hours
* Any cardiac pathology (valvulopathy, angina, ventricular arrhythmia or atrial fibrillation), vascular (arteritis obliterating the lower limbs, stenosis of the arteries with encephalic destiny, coronary artery disease) or significant respiratory (asthma, Chronic obstructive pulmonary disease, interstitial pathology)
* Alcohol consumption within 8 hours
* Ophthalmoparesis or incapacitating nystagmus (impossibility of correctly evaluating the fundus)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-22 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
To compare the wall / lumen ratio (WLR) of retinal arterioles (common marker of microangiopathies) between multiple sclerosis patients and controls using the adaptive optics technique. | Day 0

SECONDARY OUTCOMES:
Compare between patients with multiple sclerosis and controls, retinal arteriolar gauges measured by external and internal diameter. | Day 0
Correlate possible changes in arteriolar WLR with internal and external diameter, smoking, age, blood pressure, fatigue (MFIS), cognition (MDT) and disability (EDSS) scores to ambient air and normobaric oxygen. | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- CH de Versailles, Le Chesnay, France